CLINICAL TRIAL: NCT04312594
Title: A Multicenter, Randomized, Double-Blind,Placebo-controlled,Phase 2 Study of Jaktinib Hydrochloride Tablets in Participants With Idiopathic Pulmonary Fibrosis
Brief Title: Study of Jaktinib Hydrochloride Tablets in Participants With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAK005
Record Dates: First submitted 2020-02-27; First posted 2020-03-18 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jaktinib 50mg BID (Experimental): Patients receive the dose of Jaktinib Hydrochloride Tablets orally 50mg twice daily (BID) for 24 weeks.
  Interventions: Drug: Jaktinib Hydrochloride Tablets
- Jaktinib 75mg BID (Experimental): Patients receive the dose of Jaktinib Hydrochloride Tablets orally 75mg twice daily (BID) for 24 weeks.
  Interventions: Drug: Jaktinib Hydrochloride Tablets
- Placebo (Placebo Comparator): Patients receive the dose of placebo orally twice daily (BID) for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablets — Patients were administered Jaktinib taken orally as tablets twice daily
  Other Names: Jaktinib
  Arms: Jaktinib 50mg BID
Drug: Jaktinib Hydrochloride Tablets — Patients were administered Jaktinib taken orally as tablets twice daily
  Other Names: Jaktinib
  Arms: Jaktinib 75mg BID
Drug: Placebo — Patients were administered Placebo taken orally as tablets twice daily
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blinded, and placebo-controlled phase II study to evaluate the efficacy and safety of Jaktinib Hydrochloride Tablets in Participants With Idiopathic Pulmonary Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed;at least 50 years of age;no gender limitation.
2. Diagnosed idiopathic pulmonary fibrosis(see 2018.9 guidance that AST and ERS and JRS and ALAT publish );
3. FVC%≥45% normal predicted value;
4. DLCO≥30% normal predicted value；
5. FEV1 / FVC ≥0.7

Exclusion Criteria:

1. A plan of lung transplant after into group for one year.
2. In addition of IPF,Other causes cause interstitial lung disease in patients；
3. Patients with bleeding tendency (INR > 2, PT or APTT > 1.5 times normal) or cerebral hemorrhage in the past 1 year;
4. Have used anticoagulant drugs within 1 month（Except for low molecular weight heparin）;
5. An alcoholic or drug abuser;
6. Expected survival ≤ one year;
7. Patients who plan to undergo a operation within study period, such as major operations on chest and abdomen;
8. Previous use of a JAK inhibitor for more than 10 days or treatment failure;
9. Suspected allergic to Jaktinib Dihydrochloride Monohydrate , similar drugs (Fedratinib,Ruxolitinib)or their excipients;
10. Patients with malignant tumors in the previous 5 years;
11. Patients with other serious diseases that investigators believe may affect patient safety or compliance;
12. Any significant clinical or laboratory abnormalities that the investigator considers to affect safety assessment, such as: a. uncontrolled diabetes (13.9 tendency > / L), b. had high blood pressure and antihypertensive drug treatment under two or unable to descend to the ranges (systolic blood pressure < 160 mmHg, diastolic pressure < 100 mmHg), c. peripheral neuropathy (NCI - CTC AE v5.0 standard grade 2 or above)；
13. Patients hospitalized for deterioration or acute exacerbation of IPF within 1 month prior to screening;
14. patients who had not fully recovered from surgery within 1 month prior to screening;
15. Participate in clinical trials of other new drugs or medical devices within 3 months before screening;
16. Prednisone > 15mg/ day or equivalent within 1 month prior to screening;
17. Those who had used pirfenidone, Nintedanib, azathioprine, cyclophosphamide, cyclosporine A or other immunosuppressive drugs within 1 month prior to screening;
18. A history of congestive heart failure, uncontrolled or unstable angina or myocardial infarction, cerebrovascular accident or pulmonary embolism occurred within 6 month prior to screening;
19. Patients with active TB in the 12 months prior to screening;
20. Screening patients with arrhythmia requiring treatment, or with QTcB >480ms;
21. At the time of screening, there was evidence of severe impairment of organ function : including ALT and AST > 2.5uln;DBIL and TBIL > 2.0 ULN;Serum creatinine > was 1.5 ULN.
22. Evidence of active and uncontrolled viral infections such as HIV, HBV (HBsAg positive, hbv-dna positive or ≥10000 copies /ml), HCV (anti-hcv antibody or hcv-rna positive), or bacterial, viral, parasitic or fungal infections requiring treatment with any clinical symptoms;
23. patients with a history of progressive multifocal leukoencephalopathy in Screening ;
24. Patients with epilepsy or using antipsychotics(Sleep medicine,for diazepam expect) for treatment of mental illness( schizophrenia,depressed,mania,anxiety,and so on) at the time of screening;
25. Women who are planning to become pregnant or who are pregnant or breast-feeding and who are unable to use effective contraception throughout the trial period;Male patients who did not use condoms during administration and within 1 month after the last dose;
26. Subjects who cannot be treated and followed up according to the protocol;
27. Any subject whom the investigator considers inappropriate for this clinical study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Changes in forced vital capacity (FVC) [ Time Frame: 24 weeks ] | 24 weeks
  Changes in FVC from 24 weeks to baseline

SECONDARY OUTCOMES:
Progression-free time [ Time Frame: the onset of disease or death from any cause ] | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  The time from a random date to the onset of disease or death from any cause;
Non-worsening survival time: [ Time Frame:the time from randomization to the first acute exacerbation ]; | from randomization to one month
  acute aggravation events should meet all the following conditions: (1) acute exacerbation or aggravation of respiratory distress within 1 month;Chest CT showed new bilateral ground glass shadows or pulmonary interstitial fibrosis with pulmonary consolidation;(3) exclude heart failure, fluid retention and infection caused by acute dyspnea
K-BILD Scale: absolute value of change from baseline [ Time Frame: 24 weeks ] | 24 weeks
  absolute value of change from baseline at 24 weeks
mMRC Dyspnea scale：absolute value of change from baseline [ Time Frame: 24 weeks ] | 24 weeks
  absolute value of change from baseline at 24 weeks
Survival rate: [ Time Frame: 6 months, 12 months, 24 months ] | 6 months, 12 months, 24 months
  Survival rate
The severity and incidence of all adverse events and adverse reactions[ Time Frame: within 28 days after the signing of the informed consent] | within 28 days after the signing of the informed consent
  The severity and incidence of all adverse events and adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China